CLINICAL TRIAL: NCT07018323
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2b Study to Assess the Efficacy, Safety, and Tolerability of IMVT-1402 as Treatment for Adult Patients With Graves' Disease
Brief Title: A Study to Assess the Efficacy, Safety, and Tolerability of IMVT-1402 as Treatment for Adult Participants With Graves' Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMVT-1402-2503; 2025-521920-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-14; First posted 2025-06-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Graves' Disease
Keywords: IMVT-1402; Graves' disease; Thyroid-Stimulating Hormone Receptor; Immunoglobulin G; Antithyroid drug
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IMVT-1402 Dose 1 (Experimental)
  Interventions: Drug: IMVT-1402
- IMVT-1402 Dose 2 (Experimental)
  Interventions: Drug: IMVT-1402
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMVT-1402 — Dose 1 for 26 weeks
  Arms: IMVT-1402 Dose 1
Drug: IMVT-1402 — Dose 2 for 26 weeks
  Arms: IMVT-1402 Dose 2
Drug: Placebo — For 26 weeks
  Arms: Placebo

SUMMARY:
This is a multi-center, global, randomized, double-blind, placebo-controlled Phase 2b study to assess the efficacy, safety, and tolerability of IMVT-1402 in adult participants with Graves' disease (GD) who are hyperthyroid despite antithyroid drug (ATD) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the ability to understand the requirements of the trial, provide written informed consent, and comply with the trial protocol procedures.
* Male or female participants aged ≥ 18 years.
* Participants with diagnosis of GD who are hyperthyroid despite ATD treatment.
* Other, more specific inclusion criteria are defined in the protocol.

Exclusion Criteria:

* Have previously been successfully treated with radioactive iodine (RAI) therapy or have undergone total thyroidectomy.
* Have an autoimmune disease other than GD requiring treatment that, in the Investigator's judgment, puts the participant at undue risk.
* Have moderate-to-severe active thyroid eye disease (TED) and are expected to require immediate surgical intervention and/or are planning corrective surgery/irradiation or medical therapy for TED during study participation.
* Additional exclusion criteria are defined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who are euthyroid and off ATD at Week 26 (Dose 1) | Week 26

SECONDARY OUTCOMES:
Percentage of participants who have triiodothyronine (T3) (Total of T3 or free triiodothyronine [FT3]) and free thyroxine (FT4) ≤ upper limit of normal (ULN) and are off ATD at Week 26 (Dose 1) | Week 26
Percentage of participants who are euthyroid, off ATD, and seronegative at Week 26 (Dose 1) | Week 26
Percentage of participants who are euthyroid and off ATD at Week 26 (Dose 2) | Week 26
Percentage of participants who have T3 (Total T3 or FT3) and FT4 ≤ ULN and are off ATD at Week 26 (Dose 2) | Week 26
Percentage of participants who are euthyroid, off ATD, and seronegative (Dose 2) | Week 26
Percentage of participants who have T3 (Total T3 or FT3) and FT4 ≤ ULN at Week 4 in participants who have T3 (Total T3 or FT3) and/or FT4 > ULN at baseline (Dose 1) | Baseline, Week 4
Percentage of participants who have T3 (Total T3 or FT3) and FT4 ≤ ULN at Week 2 in participants who have T3 (Total T3 or FT3) and/or FT4 > ULN at baseline (Dose 1) | Baseline, Week 2
Percentage of participants who have T3 (Total T3 or FT3) and FT4 ≤ ULN at Week 4 in participants who have T3 (Total T3 or FT3) and/or FT4 > ULN at baseline (Dose 2) | Baseline, Week 4
Percentage of participants who have T3 (Total T3 or FT3) and FT4 ≤ ULN at Week 2 in participants who have T3 (Total T3 or FT3) and/or FT4 > ULN at baseline (Dose 2) | Baseline, Week 2

CONTACTS AND LOCATIONS:
Locations (97):
- United States (32):
  - Site Number - 1015, Tucson, Arizona
  - Site Number -1014, Concord, California
  - Site Number - 1013, Aurora, Colorado
  - Site Number - 1024, Doral, Florida
  - Site Number - 1008, Hialeah, Florida
  - Site Number - 1000, Miami, Florida
  - Site Number - 1020, Columbus, Georgia
  - Site Number - 1022, Topeka, Kansas
  - Site Number - 1033, Jefferson City, Missouri
  - Site Number - 1004, Kansas City, Missouri
  - Site Number - 1019, St Louis, Missouri
  - Site Number - 1012, Reno, Nevada
  - Site Number - 1032, Long Island City, New York
  - Site Number - 1027, New Hyde Park, New York
  - Site Number - 1009, New York, New York
  - Site Number - 1018, Williamsville, New York
  - Site Number - 1010, Chapel Hill, North Carolina
  - Site Number - 1026, Hickory, North Carolina
  - Site Number - 1001, Morehead City, North Carolina
  - Site Number - 1034, Raleigh, North Carolina
  - Site Number - 1007, Oklahoma City, Oklahoma
  - Site Number - 1017, Memphis, Tennessee
  - Site Number - 1029, Dallas, Texas
  - Site Number - 1002, El Paso, Texas
  - Site Number - 1003, Fort Worth, Texas
  - Site Number - 1031, Houston, Texas
  - Site Number - 1028, Houston, Texas
  - Site Number -1023, Irving, Texas
  - Site Number - 1021, Irving, Texas
  - Site Number - 1025, McKinney, Texas
  - Site Number - 1011, San Antonio, Texas
  - Site Number - 1016, Norfolk, Virginia
- Australia (7):
  - Site Number - 5105, Sydney, New South Wales
  - Site Number - 5103, Warrawong, New South Wales
  - Site Number - 5101, Brisbane, Queensland
  - Site Number - 5100, Southport, Queensland
  - Site Number - 5104, Geelong, Victoria
  - Site Number - 5108, Perth
  - Site Number - 5109, Saint Leonards
- Bulgaria (12):
  - Site Number - 5613, Dobrich
  - Site Number - 5606, Plovdiv
  - Site Number - 5607, Plovdiv
  - Site Number - 5601, Sliven
  - Site Number - 5612, Smolyan
  - Site Number - 5604, Sofia
  - Site Number - 5609, Sofia
  - Site Number - 5608, Sofia
  - Site Number - 5602, Varna
  - Site Number - 5603, Varna
  - Site Number - 5611, Varna
  - Site Number - 5600, Yambol
- Czechia (4):
  - Site Number - 3203, Náchod
  - Site Number - 3201, Prague
  - Site Number - 3200, Prague
  - Site Number - 3202, Prague
- Georgia (6):
  - Site Number - 8004, Imereti
  - Site Number - 8003, Tbilisi
  - Site Number - 8000, Tbilisi
  - Site Number - 8002, Tbilisi
  - Site Number - 8001, Tbilisi
  - Site Number - 8005, Tbilisi
- Greece (3):
  - Site Number - 3902, Athens
  - Site Number - 3900, Athens
  - Site Number - 3901, Athens
- Israel (10):
  - Site Number - 4202, Ramat Gan, Central District
  - Site Number - 4205, Haifa, Haifa District
  - Site Number - 4203, Haifa, Haifa District
  - Site Number - 4209, Nahariya, Northern District
  - Site Number - 4206, Tzfat, Northern District
  - Site Number - 4211, Beersheba, Southern District
  - Site Number - 4201, Jerusalem
  - Site Number - 4204, Jerusalem
  - Site Number - 4200, Petah Tikva
  - Site Number - 4207, Tel Aviv
- Latvia (5):
  - Site Number - 4600, Ogre
  - Site Number - 4602, Riga
  - Site Number - 4603, Riga
  - Site Number - 4604, Sigulda
  - Site Number - 4601, Ventspils
- New Zealand (2):
  - Site Number - 3301, Auckland
  - Site Number - 3300, Wellington
- Poland (8):
  - Site Number - 3002, Bydgoszcz
  - Site Number - 3010, Chorzów
  - Site Number - 3007, Kielce
  - Site Number - 3000, Lublin
  - Site Number - 3005, Olsztyn
  - Site Number - 3009, Opole
  - Site Number - 3006, Poznan
  - Site Number - 3008, Warsaw
- South Korea (6):
  - Site Number - 4500, Daegu
  - Site Number - 4503, Goyang
  - Site Number - 4504, Guri-si
  - Site Number - 4501, Seoul
  - Site Number - 4506, Seoul
  - Site Number - 4505, Seoul
- United Kingdom (2):
  - Site Number - 7009, Cornwell
  - Site Number - 7001, London

IPD SHARING:
Plan to Share IPD: No